CLINICAL TRIAL: NCT05813041
Title: A Single-site, First-in-human Trial to Assess the Safety and Performance of a Novel Device, the BioCaptis, for Capturing Cell-free DNA (cfDNA) in Healthy Human Subjects When Used in an Apheresis Circuit
Brief Title: A First-in-human Trial to Assess the Safety and Performance of the BioCaptis in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioCaptiva Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BioCaptis-1
Record Dates: First submitted 2023-01-11; First posted 2023-04-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Clinical investigation of the safety and performance of a medical device. Single site, single arm, open label, healthy volunteer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Device (Experimental): Single arm trial - healthy volunteers will all undergo an apheresis procedure using the BioCaptis device. No comparator will be used for this trial.
  Interventions: Device: BioCaptis

INTERVENTIONS:
Device: BioCaptis — The BioCaptis is a medical device intended to capture cell-free DNA from peripheral blood for use in liquid biopsy. When used as a cartridge filter during an apheresis procedure in which plasma is passed through the device, the BioCaptis binds cfDNA which can be eluted, concentrated, and used as an input for cancer diagnostic tests.

SUMMARY:
Liquid biopsy is a new field in medicine where doctors can look at small molecules in our blood, called DNA, that carry the genetic material that makes us who we are. In some illnesses this DNA starts behaving abnormally, meaning that these illnesses can be identified by looking closely at changes in a person's DNA.

The BioCaptis is a new medical device which can capture molecules of DNA, called cell-free DNA, from a person's blood when used in a clinical procedure called apheresis. The purpose of the BioCaptis-1 clinical trial is to confirm that the BioCaptis is suitable for use in healthy volunteers. The main questions the study aims to answer are:

* Is the BioCaptis safe to use in healthy volunteers?
* Can the BioCaptis capture cell-free DNA from human plasma when used in an apheresis procedure?

Following completion of the informed consent process, participants in the study will complete six appointments over the course of the trial. Three of these will be telephone appointments, and three will be in-person visits at the clinical site. The three in-person visits will include:

* Screening Visit where screening tests will be performed to deem the participant suitable for enrollment;
* Procedural Visit during which the participant will undergo the apheresis procedure with the BioCaptis device;
* Post-procedure Follow Up Visit to check the particpant's health following the apheresis procedure.

DETAILED DESCRIPTION:
Personalised medicine is a medical model which has developed rapidly in recent years, and it involves tailoring treatment plans to individual patients based on the type of disease they have and how they are expected to respond to certain treatment types. To develop personalised treatment plans for cancer patients, doctors look at a piece of tumour tissue taken from the patient which is called a biopsy. Doctors will examine this biopsy to identify genetic abnormalities which help to explain the behaviour of that tumour or indicate how that tumour could respond to certain anti-cancer treatments. This is called "molecular profiling."

Although tissue biopsy is widely used for molecular profiling, it has some drawbacks. Firstly, tissue biopsy is a highly invasive procedure which can cause stress to patients. Secondly, some biopsies are performed using a small needle, and due to the small size of this needle the tumour tissue can be missed meaning that there is no tumour tissue present in the sample to carry out necessary tests. Thirdly, tissue biopsy can't be used for real-time monitoring of cancers because multiple biopsies would be required from a patient over the course of their treatment which would cause additional stress and discomfort to them. So, an alternative biopsy method is needed to address these limitations.

A new field in medicine called "liquid biopsy" is becoming very popular. This is where a doctor can use a blood sample to diagnose an illness instead of having to take a tissue biopsy. Liquid biopsy works by looking at very small molecules in our blood, called DNA, that carry the genetic material that makes us who we are. In some illnesses this DNA starts behaving abnormally, meaning that these illnesses can be identified by looking closely at a person's DNA. One illness that liquid biopsy has the potential to identify is cancer because DNA from all the body's cells, including cancer cells, can be found in the blood stream. Doctors can then use this information to choose a treatment plan for the patient. Although it shows promise for use in molecular profiling, development of liquid biopsy has been held back because the amount of DNA that can be collected using a regular blood draw (the kind used in a doctor's surgery) is very low and does not give reliable results when used in laboratory tests. To address this limitation, BIOCAPTIVA has developed a medical device called the BioCaptis which is a small tube that has a special filter in it. The filter can capture up to 100 times more cfDNA than a regular blood sample when it is used during an apheresis procedure.

An apheresis procedure is a routine and safe process used to treat patients with a range of conditions. It is also used to collect blood cells from healthy donors that can then be used to treat sick patients. It works by connecting a patient or healthy donor to a machine. Blood flows from the person into the machine where it is then separated out into its main parts. The part of the blood that is causing the patient's condition, or contains the cells that can be used to treat patients, is removed and everything else is returned back to the person. Apheresis is a well-tolerated procedure, but as with all procedures there is some risk. The most commonly observed side effects are listed below:

* Bruising can occur at the needle puncture site.
* Sometimes the blood vessel that the needle has been placed in goes into spasm, so the blood flow slows down.
* A blood thinner is added into the machine to stop the person's blood from clotting while it is outside of their system. Some of it flows back into their system with the blood being returned which can cause tingling around the mouth or fingertips, or cause shivering.

The BioCaptis-1 study has been designed to confirm that the BioCaptis device is both safe to use and able to capture DNA from the blood of human subjects when used with an apheresis procedure. In this clinical trial, we will use an apheresis machine in combination with the BioCaptis device. The participant's plasma will pass through the BioCaptis and the filter inside the device will capture the DNA in the participant's plasma. Their plasma will then be combined with the rest of their blood and be returned to them.

As this is a completely new device, no similar research on this topic has been done before.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study
* All genders aged 18-60 years (inclusive)
* Healthy volunteer study therefore subjects must be deemed to be in good health by the Investigator
* Subject has acceptable clinical history at point of enrolment
* Subject has clinically acceptable laboratory and ECG assessments at point of enrolment
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow their General Practitioner (and all other relevant healthcare providers as appropriate) to be notified of participation in the study
* Adequate bilateral peripheral venous access (antecubital fossae, forearms) for apheresis catheter placement.

Exclusion Criteria:

* Subjects who are pregnant, lactating or planning pregnancy during the study
* Significant renal or hepatic impairment, or any disorder of blood cells or of blood coagulation
* Scheduled elective surgery, or other procedures requiring general anaesthesia, during the subject's time enrolled in the study
* Any significant disease or disorder, or any regular drug treatments which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study
* Donation of blood within the 12 weeks prior to enrolment
* Donation of platelets within the 3 weeks prior to enrolment
* Subjects who have participated in another research study involving an investigational product in the past 12 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The adverse events profile observed for all participants undergoing the investigational procedure to evaluate the safety of the BioCaptis device. | Up to 7 days post-procedure
  To assess the safety of the BioCaptis device as a binding column in an apheresis circuit in healthy human subjects. The outcome measure will be the adverse event profile (i.e. adverse device effects and serious adverse device effects) observed for healthy human subjects undergoing an apheresis procedure using the BioCaptis device.
The amount of cfDNA (nanograms) that can be eluted and concentrated from the BioCaptis device after use to evaluate the performance of the device. | Immediately after the procedure
  To confirm that the BioCaptis device can capture cfDNA, when used in an apheresis circuit. The outcome measure will be the amount of cfDNA (nanograms) that can be eluted and concentrated from the BioCaptis device after use of the device in an apheresis procedure.

SECONDARY OUTCOMES:
For each subject, measure the amount of cfDNA collected using the BioCaptis device and compare it with the amount of cfDNA obtained from a paired 10mL blood draw in healthy human subjects | Immediately after the procedure
  The amount of cfDNA obtained using the BioCaptis and from a paired 10mL blood draw.
For each subject, assess the fragment size profile of cfDNA collected using the BioCaptis and compare it with cfDNA obtained from a paired 10mL blood draw. | Immediately after the procedure
  The fragment size distribution of cfDNA obtained using the BioCaptis and from a paired 10mL blood draw.
For each subject, assess the performance in molecular genetic assays, such as qPCR, of cfDNA obtained using the BioCaptis device and compare it with the performance of cfDNA obtained from a paired 10mL blood draw. | Up to 7 days post-procedure
  The amplification efficiency in a qPCR assay of cfDNA captured using the BioCaptis device and from a paired 10mL blood draw.

IPD SHARING:
Plan to Share IPD: No